CLINICAL TRIAL: NCT00734279
Title: Follicle-Stimulating Hormone (FSH) and the Onset of Puberty
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Michigan (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Carol Foster, Professor, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-3125; 5M01RR000064 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-08-14 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Delayed Puberty; Precocious Puberty
Keywords: Puberty; Delayed; Early; Precocious; Peripubertal; Gonadotropin; FSH; LH
MeSH Terms: conditions — Puberty, Delayed; Puberty, Precocious | interventions — Leuprolide; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Girls with Early Puberty receive ganirelix and leuprolide acetate to determine effect of ganirelix on gonadotropin secretion
  Interventions: Drug: Leuprolide Acetate - Early Puberty Leuprolide Visit; Drug: Ganirelix - Early Puberty Ganirelix Visit
- 2 (Experimental): Girls with Delayed Puberty receive ganirelix and leuprolide acetate to determine effect of ganirelix on gonadotropin secretion
  Interventions: Drug: Ganirelix - Delayed Puberty Ganirelix Visit; Drug: Leuprolide Acetate- Delayed Puberty Leuprolide Visit
- 3 (Experimental): Boys with Early Puberty receive ganirelix and leuprolide acetate to determine effect of ganirelix on gonadotropin secretion
  Interventions: Drug: Leuprolide Acetate - Early Puberty Leuprolide Visit; Drug: Ganirelix - Early Puberty Ganirelix Visit
- 4 (Experimental): Boys with Delayed Puberty receive ganirelix and leuprolide acetate to determine effect of ganirelix on gonadotropin secretion
  Interventions: Drug: Ganirelix - Delayed Puberty Ganirelix Visit; Drug: Leuprolide Acetate- Delayed Puberty Leuprolide Visit

INTERVENTIONS:
Drug: Leuprolide Acetate - Early Puberty Leuprolide Visit — Dose of 10 mcg/kg Sub cutaneous once at 0800 on day 2 of the Early Puberty Luprolide Visit
  Other Names: Leuprolide Injection; Lupron; Lupron SQ; Lupron Injection; Leuprolide SQ
  Arms: 1; 3
Drug: Ganirelix - Early Puberty Ganirelix Visit — Dose of 2.5 mcg/kg Sub-cutaneous once at 17:30 on day 1 of the Early Puberty Ganirelix Visit and once at 08:00 on day 2 of the Early Puberty Ganirelix Visit
  Other Names: Ganirelix SQ; Ganirelix Acetate
  Arms: 1; 3
Drug: Ganirelix - Delayed Puberty Ganirelix Visit — Ganirelix is administered at a dose of 2.5 mcg/kg sub cutaneous at 17:30 on day 1 and once at 08:00 on day 2 of the Ganirelix Delayed Puberty Visit
  Other Names: Ganirelix SQ; Ganirelix Acetate
  Arms: 2; 4
Drug: Leuprolide Acetate- Delayed Puberty Leuprolide Visit — Leuprolide acetate is given at a dose of10 mcg/kg at 0800 on day 2 of the Delayed Puberty Leuprolide Visit
  Other Names: Leuprolide Injection; Lupron; Lupron SQ; Lupron Injection; Leuprolide SQ
  Arms: 2; 4

SUMMARY:
The purpose of this study is to determine if the timing of the onset of puberty may be affected by FSH-regulatory peptides.

We will determine how these peptides relate to FSH production in prepubertal and pubertal children by comparing the regulation of FSH control in children with precocious (early) puberty and delayed puberty.

In this pilot study, we will stimulate the pubertal axis using an agonist of GnRH to determine the pubertal response of activin-A, inhibin-A and -B and follistatin.

To determine baseline FSH secretion and FSH-regulatory peptide tone, we will block GnRH with a specific antagonist.

These studies should lead to a better understanding of the role of FSH in controlling the onset of puberty and the pathogenesis of pubertal disorders.

DETAILED DESCRIPTION:
Girls begin puberty earlier and have as much as a 5-fold increase in incidence of precocious puberty as do boys, while boys are more likely to have delayed adolescence compared to girls.

The reasons for sex differences in the timing of puberty and sex-based variation in expression of pubertal disorders are not known.

Puberty is heralded by an increase in the episodic release of luteinizing hormone (LH) under the control of increased gonadotropin-releasing hormone (GnRH) release. It has been thought that sex differences in central nervous system restraint of GnRH and subsequently of LH secretion account for the differences in timing of onset of puberty in boys and girls.

Follicle-stimulating hormone (FSH) secretion is readily detected prior to the onset of puberty and exhibits sexual dimorphism in basal and GnRH-stimulated concentrations. Thus, assessment of factors regulating FSH secretion during childhood may enhance our understanding of sex differences in pubertal development and the pathogenesis of precocious puberty.

Although FSH is secreted under the control of GnRH, FSH is also secreted constitutively under the control of a group of peptides collectively known as the FSH-regulatory proteins. These peptides include activins, peptides that increase FSH secretion and inhibins and follistatins, peptides that suppress FSH secretion.

Gonadal inhibins inhibit FSH via endocrine negative feedback, but their production during puberty is only beginning to be understood. Activin and follistatin have been thought to have a principle paracrine role in FSH regulation but recent data have demonstrated these peptides have an endocrine role as well.

We hypothesize that differences in elaboration of activins, inhibins, and follistatin that alter FSH constitutive secretion underlie precocious and delayed puberty in boys and girls and account, in part, for sex differences in pubertal timing.

Specifically we expect that the inhibitory regulators, inhibins and/or follistatins, will be lower while the stimulatory regulator, activin, will be higher in early compared to delayed puberty.

FSH and the Onset of Puberty is a case control study comparing boys with precocious puberty to boys with delayed adolescence and girls with precocious puberty to girls with delayed adolescence.

Hypothesis: Basal and GnRH agonist-stimulated activin concentrations will be greater and inhibin concentrations lower in children with early puberty than in children with delayed adolescence, and the GnRH antagonist, ganirelix, will decrease activin concentrations in children with early puberty but not in delayed adolescence.

Specific Aim 1: Determine the degree to which FSH-regulatory peptides, compared to gonadotropin-releasing hormone (GnRH), control FSH secretion in children by suppressing GnRH with ganirelix in children with early and delayed adolescence.

Specific Aim 2: Determine the role of FSH-regulatory peptides in control of timing of onset of puberty by comparing their concentrations with and without GnRH stimulation of FSH in children with precocious puberty and delayed adolescence.

Specific Aim 3: Determine the role of GnRH in control of the FSH-regulatory peptides by comparing activin, inhibin and follistatin concentrations in children with delayed adolescence due to constitutional growth delay to those with delayed adolescence from hypogonadotropic hypogonadism

ELIGIBILITY:
Inclusion Criteria:

Early Puberty Children who have early puberty may participate in this study. Children must be between 6 and 10 years of age and be healthy with the exception of having early puberty. For early puberty, girls should have had the onset of breast development prior to 8 years of age and boys should have the onset of pubic hair growth or genital growth prior to 9 years of age.

Inclusion Criteria for Delayed Puberty Children who have late (delayed) puberty may participate in this study. Children must be between 12 and 17 years of age and be healthy with the exception of having late puberty. In order to have late puberty, boys and girls should have short stature compared to their family with at least one year delay in bone age as determined by bone age x-ray and/or have the onset of secondary sexual characteristics (breast and pubic hair growth) at 12 years of age or later for a girl or 13 years of age or later for a boy.

Exclusion Criteria:

Early Puberty Children with known genetic disorders, chronic medical conditions requiring the use of steroids, and use of medication for puberty within the last 3 months are excluded.

Delayed Puberty Children with known genetic disorders with the exception of possible hypogonadotropic hypogonadism, chronic medical conditions requiring the use of steroids, and use of medication for puberty within the last 3 months are excluded.

-

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2006-03; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Determine the ability of the GnRH antagonist, ganirelix, to suppress nocturnal gonadotropin secretion in peripubertal boys and girls | Sample analysis is conducted after the leuprolide portion of the study and the ganirelix portion of the study have been completed for the first 6 patients

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Foster, MD, Principal Investigator — University of Utah, Department of Pediatric Endocrinology
Locations (1):
- Utah Diabetes Center, Salt Lake City, Utah, United States